CLINICAL TRIAL: NCT02004782
Title: Reduction in Symptomatic Oesophageal Stricture Formation Post-two Stage Complete Barrett's Excision for High Grade Dysplasia or Early Adenocarcinoma With Short-term Steroid Therapy: A Randomized, Doubleblind, Placebo-controlled, Multicentre Trial.
Brief Title: Barretts oEsophageal Resection With Steroid Therapy Trial
Acronym: BERST
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: study abandoned
Sponsor: Professor Michael Bourke (Other)
Responsible Party: Sponsor-Investigator, Professor Michael Bourke, Professor, Western Sydney Local Health District
Organization: Western Sydney Local Health District (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: HREC2013/7/4.5(3702)
Record Dates: First submitted 2013-11-25; First posted 2013-12-09 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Barrett Esophagus; Esophageal Stenosis
MeSH Terms: conditions — Barrett Esophagus; Esophageal Stenosis | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prenisolone (Active Comparator): Daily prednisolone is taken for 6 weeks, at a dose of 40mg in week 1, 30mg in week 2, 20mg week 3 and 4, 10mg in week 5, and 5mg in week 6. Prednisolone is taken in the morning. Treatment commences the day of the procedure, with the dose taken with a sip of water prior to discharge. The 6-week treatment regimen is given after both the 1st and 2nd stage CBE.
  Interventions: Drug: Prednisolone
- Placebo (Placebo Comparator): Daily placebo is taken for 6 weeks, at a dose of 40mg in week 1, 30mg in week 2, 20mg week 3 and 4, 10mg in week 5, and 5mg in week 6. Placebo is taken in the morning. Treatment commences the day of the procedure, with the dose taken with a sip of water prior to discharge. The 6-week treatment regimen is given after both the 1st and 2nd stage CBE.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Prednisolone — Daily prednisolone is taken for 6 weeks, at a dose of 40mg in week 1, 30mg in week 2, 20mg week 3 and 4, 10mg in week 5, and 5mg in week 6. Prednisolone is taken in the morning. Treatment commences the day of the procedure, with the dose taken with a sip of water prior to discharge. The 6-week treatment regimen is given after both the 1st and 2nd stage CBE.
  Arms: Prenisolone
Drug: Placebo Oral Tablet — Daily placebo is taken for 6 weeks, at a dose of 40mg in week 1, 30mg in week 2, 20mg week 3 and 4, 10mg in week 5, and 5mg in week 6. Placebo is taken in the morning. Treatment commences the day of the procedure, with the dose taken with a sip of water prior to discharge. The 6-week treatment regimen is given after both the 1st and 2nd stage CBE
  Arms: Placebo

SUMMARY:
Barretts mucosa is a premalignant condition of the oesophagus, which can progress to cancer. Oesophageal cancer is aggressive, with a 5 year survival of only ~15%. High risk Barretts mucosa, containing high grade dysplasia or early cancer, can be removed by endoscopic mucosal resection (EMR) during gastroscopy. If patients can be effectively treated by EMR while they have premalignant or early malignant disease, it is a curative procedure.

Currently, the major limitation of Complete Barretts Excision (CBE) by EMR, is scar tissue development in the oesophagus, leading to stricture formation and difficulty swallowing (dysphagia). If a safe and effective method could be found to reduce this risk, the treatment options for early oesophageal cancer would be greatly improved. CBE is performed as a two stage procedure, with 2 gastroscopies 8 weeks apart. In this randomised, doubleblind study, eligible and enrolled patients are randomised after the 1st stage CBE to receive either prednisolone tablets or placebo. Inclusion criteria are patients with short segment (<3cm circumferential disease) Barretts oesophagus with high grade dysplasia or early cancer. The treatment period is for 6 weeks after both CBE sessions. Prednisolone is given in a reducing dose over the 6 weeks, starting at 40mg daily.

The primary outcome is symptomatic dysphagia development. Endoscopic dilation will be performed as required for dysphagia secondary to symptomatic oesophageal stricture formation persisting for ≥2 days, or complete dysphagia for any time period. Endoscopic surveillance with biopsies will occur at a 3 month, 6 month then 12 month interval following CBE, to assess for complete removal of Barretts mucosa.

Following two stage CBE, stricture rates without preemptive therapy in noncircumferential, circumferential <2cm, and circumferential <3cm disease, are estimated to be 30%, 50% and 70% respectively. The investigators predict a 50% reduction in stricture rate with oral steroid therapy. With a primary analyses of oral steroid versus placebo tested at a 5% level of significance in a two tailed test, 58 patients are needed per group. Allowing for a 5% drop out rate, a total of 126 patients are required. The study will be performed at five Australian Tertiary Hospitals, and the recruitment period is estimated to be 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed Barretts mucosa with High Grade Dysplasia or early adenocarcinoma (T1a, intramucosal adenocarcinoma).
2. Barretts segment ≥ 30% circumference, ≤C3 and ≤M5.
3. The general health condition of the patient permits anaesthesia for endoscopy.
4. Patient is 18 years of age or older.
5. Informed consent is obtained

Exclusion Criteria:

1. Previous (referral) biopsies show low grade dysplasia only, or invasive adenocarcinoma.
2. Barretts segment <30% circumference, >C3 or >M5.

4. During initial gastroscopy there are highly suspicious areas for submucosal invasive cancer (Kudo pit pattern type V; excavated/depressed type morphology; large smooth or ulcerated nodule). In cases of significant doubt, initial resection is of the highly suspicious area only, and urgent histology processing requested. If submucosal invasion is excluded, the patient is rebooked for 1st stage CBE (60% circumferential resection) and randomization after a 4-6 weeks interval.

4. Presence of a tight peptic oesophageal stricture that impedes safe and effective EMR using the Duette cap.

5. Active malignancy, uncontrolled Diabetes Mellitus, active or untreated major psychiatric disorder, uncontrolled infection, uncontrolled hypertension, uncontrolled or severe congestive cardiac failure, non-correctable coagulopathy (INR>2, or platelet count <60 x 109/L), osteoporosis, recent peptic ulcer disease, moderate-to-severe glaucoma or untreated glaucoma, or pregnancy.

6. Unable to provide informed consent 7. Allergy to compound used in tablet formulation: Microcrystalline cellulose (MCC).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Rate of symptomatic stricture formation | >2 days
  Rate of symptomatic oesophageal stricture formation.A symptomatic stricture is defined as a stricture leading to the inability to tolerate a soft diet for ≥ 2 days, or the presence of complete dysphagia for any length of time.

SECONDARY OUTCOMES:
Dilations | Two weeks or more
  The need for, and number of endoscopic dilations.
Dysphagia score | 3, 6 and 12 months
  Dysphagia score (DS) at 3, 6 and 12 month surveillance endoscopies. DS: 0 = Normal diet; 1 = Some solid foods; 2 = Semi-solid foods; 3 = Liquids only; 4 = Total dysphagia
Stricture formation | 3, 6, 12 months
  Endoscopic evidence of stricture formation at 3, 6 and 12 month surveillance endoscopies. No stricture, mild stricture, moderate stricture ('hugs' the gastroscope but the gastroscope can pass), severe stricture (cannot be passed with the gastroscope)
Recurrence | 3, 6 and 12 months
  Recurrence of Barretts mucosa, defined as the presence of Barretts mucosa endoscopically, or mucosal columnar epithelium with or without intestinal metaplasia on surveillance biopsies. Measured at 3-month surveillance (20 weeks post 1st CBE), 6 month surveillance (46 weeks post 1st CBE), and 12 month surveillance (98 weeks post 1st CBE) endoscopies.

OTHER OUTCOMES:
Cost | 0-12 months
  The direct medical costs and indirect non-medical costs of production lost will be calculated based on Australian Medical guidelines, and compared between each treatment strategy.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bourke, Principal Investigator — Western Sydney Local Health District
Locations (1):
- Westmead Hospital, Westmead, New South Wales, Australia